CLINICAL TRIAL: NCT03127397
Title: Contribution of "Praise Messages" to HIV Treatment Retention and Adherence Among Female Sex Workers in Ethiopia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Reed College (Other)
Collaborators: Population Services International (Other); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nicholas Wilson, Associate Professor of Economics, Reed College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SERO-061-03-2017
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: HIV/AIDS
Keywords: antiretroviral therapy; HIV/AIDS; ART adherence
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention)
- Praise Message (Experimental): Receives up to two praise message phone calls after each completed ART appointment.
  Interventions: Behavioral: Praise message phone call

INTERVENTIONS:
Behavioral: Praise message phone call — Praise message phone calls after each completed ART appointment, up to two calls per month.
  Arms: Praise Message

SUMMARY:
This study evaluates the effects of praise message phone calls on antiretroviral therapy (ART) initiation, adherence, and prescription refills. The investigators will use randomization to assign newly (diagnosed) HIV positive, ART naive, female sex workers (FSWs) in Ethiopia to a praise message phone call study arm or to a standard of care control study arm.

DETAILED DESCRIPTION:
This study evaluates the effects of praise message phone calls on antiretroviral therapy (ART) initiation, adherence, and prescription refills. The investigators will use randomization to assign newly (diagnosed) HIV positive, ART naive, female sex workers (FSWs) in Ethiopia to a praise message phone call study arm or to a standard of care control study arm.

Inadequate adherence to ART medication, missed clinics visits and loss-to-follow-up, and failure to refill prescriptions are major barriers to achieving viral suppression. Non-adherence is associated with a range of individual, social, community, and structural factors, including low health literacy, a lack of social support, low socioeconomic status, substance abuse, stigma and discrimination, and a lack of access to a reliable source of ART drugs. ART patients' perceptions about a lack of health provider respect and mutual trust are a possible further barrier to adherence.

Provision of HIV therapy within the MULU/MARPs drop-in-centers has attempted to mitigate some of the structural and social barriers to ART initiation and retention in care by bringing FSW friendly treatment services closer to clients and providing intensive counseling services, social and economic support services, and referrals to additional health services. Improving client perceptions of health care provider attitudes may further improve retention in care and adherence to treatment among FSW in Ethiopia. This study will measure the effects of praise message phone calls delivered the day after, and two weeks after, completing a ART appointment (i.e. initiation and/or prescription refill) on subsequent ART refills/HIV clinic visits.

This study will be conducted within PSI/Ethiopia's USAID-funded MULU/MARPs program, which provides HIV testing, treatment, and other services to female sex workers (FSW) through a network of drop-in-centers (DICs) across Ethiopia. Consenting FSWs who are living with HIV, who are ART naive, and who are referred for ART initiation to one of the 25 drop-in-centers (DICs) selected for "Test and Start" implementation will be enrolled in the study. Pre-study analysis indicates that each DIC enrolls between 3-4 FSWs living with HIV on ART each month (mean: 3.6). Over the course of our 9 month study, the investigators expect to enroll a total of 810 study participants.

ELIGIBILITY:
Inclusion Criteria:

* Written consent,
* ART naive,
* Female sex worker,
* Living with HIV,
* And, seeking care at a participating clinic

Exclusion Criteria:

* No consent,
* Previous ART,
* Has not exchanged sex for money in past 12 months,
* HIV negative,
* And/or, has not sought care at a participating clinic

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 810 (Estimated)
Dates: Start 2017-04-20 (Actual); Primary Completion 2018-07-30 (Estimated); Study Completion 2018-07-30 (Estimated)

PRIMARY OUTCOMES:
Retention in care at 1 month | 1 month
ART adherence at 1 month | 1 month
Retention in care at 3 months | 3 months
ART adherence at 3 months | 3 months
Retention in care at 6 months | 6 months
ART adherence at 6 months | 6 months
Viral suppression at 6 months | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Addis Ababa, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: No